CLINICAL TRIAL: NCT00002499
Title: TREATMENT OF ALL IN FIRST BONE MARROW RELAPSE AFTER BFM PROTOCOLS
Brief Title: Combination Chemotherapy in Treating Children With Relapsed Acute Lymphocytic Leukemia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Grupo Argentino de Tratamiento de la Leucemia Aguda (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000077835; ARG-GATLA-1LLAREC90; NCI-F92-0006
Record Dates: First submitted 1999-11-01; First posted 2004-08-23 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2000-05

CONDITIONS: Leukemia
Keywords: recurrent childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Asparaginase; Cytarabine; Daunorubicin; Dexamethasone; Methotrexate; Prednisone; Vincristine; Radiotherapy

INTERVENTIONS:
Drug: asparaginase
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: dexamethasone
Drug: methotrexate
Drug: prednisone
Drug: vincristine sulfate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase II/III trial to study the effectiveness of combination chemotherapy in treating children with relapsed acute lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the feasibility, at GATLA, of a study of the treatment of ALL in first hematologic relapse following treatment on a BFM protocol. II. Evaluate the efficacy of induction with vincristine/daunorubicin/asparaginase/prednisone in producing a second complete remission in these patients, and evaluate the toxicity of this regimen. III. Evaluate the efficacy and toxicity of the Capizzi I regimen (vincristine/asparaginase/methotrexate) and Capizzi II regimen (cytarabine/asparaginase/daunorubicin) when given to maintain and prolong complete remission. IV. Offer the option of bone marrow transplantation to those patients who are in second remission and who have a histocompatible donor, and compare outcome of these patients with those on chemotherapy alone.

OUTLINE: Nonrandomized study. Patients achieving remission on Induction proceed to Interim Maintenance, then to Continued Maintenance; those failing to achieve remission receive Salvage Re-induction, followed, if remission is achieved, by Interim Maintenance, then Continued Maintenance. Induction: 4-Drug Combination Chemotherapy with CNS Prophylaxis/Therapy. Vincristine, VCR, NSC-67574; Prednisone, PRED, NSC-10023; Asparaginase, ASP, NSC-109229; Daunorubicin, DNR, NSC-82151; with Intrathecal Cytarabine, IT ARA-C, NSC-63878; Intrathecal Dexamethasone, IT DM, NSC-34521. Interim Maintenance: 3-Drug Combination Chemotherapy with, as indicated, Radiotherapy. VCR; ASP; Methotrexate, MTX, NSC-740; with, as indicated, testicular irradiation (equipment not specified). Continued Maintenance: 3-Drug Combination Chemotherapy followed by 3-Drug Combination Chemotherapy with CNS Prophylaxis and, as indicated, Radiotherapy. Capizzi II: ARA-C; ASP; DNR; followed by Capizzi I: VCR; ASP; MTX; with IT ARA-C; IT DM; and, as indicated, cranial irradiation (equipment not specified). Salvage Re-induction: 2-Drug Combination Chemotherapy. ARA-C; ASP.

PROJECTED ACCRUAL: At least 72 evaluable patients will be entered. Accrual is expected to be completed in 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: ALL in first hematologic relapse during or following completion of treatment on a BFM protocol (ARG-GATLA-1-LLA-82, -84, -87, or -90) M2-M3 bone marrow required

PATIENT CHARACTERISTICS: Age: Under 20 Performance status: Not specified Life expectancy: Greater than 8 weeks Hematopoietic: Not specified Hepatic: No significant liver disease Renal: No significant kidney disease Cardiovascular: No significant heart disease Pulmonary: No significant lung disease Other: No significant digestive disease

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Prior total anthracycline no greater than 280 mg/sqm Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not applicable

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1990-01

CONTACTS AND LOCATIONS:
Overall Officials: Federico Sackmann-Muriel, MD, Study Chair — Hospital de Pediatria Garrahan
Locations (1):
- Grupo Argentino de Tratamiento de la Leucemia Aguda, Buenos Aires, Buenos Aires, Argentina